CLINICAL TRIAL: NCT02592694
Title: Intracoronary Cocktail Injection Combined With Thrombus Aspiration in ST-elevation Myocardial Infarction Patients Treated With Primary Angioplasty
Brief Title: Intracoronary Cocktail Injection Combined With Thrombus Aspiration in STEMI Patients Treated With Primary Angioplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, sunddong, Principal Investigator, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cocktail I
Record Dates: First submitted 2015-10-26; First posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: ST-elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Tirofiban; bivalirudin; Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cocktail with thrombus aspiration (Experimental): Intracoronary cocktail (tirofiban, bivalirudin, tenecteplase) injection combined with thrombus aspiration
  Interventions: Drug: cocktail; Device: thrombus aspiration
- Thrombus aspiration (Active Comparator): Thrombus aspiration alone
  Interventions: Device: thrombus aspiration

INTERVENTIONS:
Drug: cocktail — Cocktail (tirofiban, bivalirudin, tenecteplase) will be given in addition to thrombus aspiration
  Other Names: tirofiban, bivalirudin, tenecteplase
  Arms: Cocktail with thrombus aspiration
Device: thrombus aspiration — manual thrombus aspiration
  Other Names: manual thrombus aspiration

SUMMARY:
This is a randomized, double blind, placebo controlled study of intracoronary cocktail injection combined with thrombus aspiration versus thrombus aspiration alone in ST-elevation myocardial infarction patients treated with primary angioplasty.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled study of intracoronary cocktail injection combined with thrombus aspiration versus thrombus aspiration alone in ST-elevation myocardial infarction patients treated with primary angioplasty. Patients with STEMI will be randomized into the cocktail group or the control group. Patients in the cocktail group will receive cocktail injection combined with thrombus aspiration. Patients in the control group will receive thrombus aspiration alone. The primary outcome of the cocktail I study is the composite of death, myocardial infarction or class IV heart failure within 1 year. The secondary outcome of the cocktail I study include slow reflow/no reflow during PCI, left ventricular function, quality of life, stroke or life-threatening bleeding within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age adult patients with STEMI Referred for primary PCI within 5d of symptom onset

Exclusion Criteria:

* Patients who had undergone previous coronary artery bypass surgery or PCI or had received fibrinolytic therapy History of stroke Active bleeding Severe hepatic or renal dysfunction Cardiogenic shock Contraindications for primary PCI or DAPT

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Death, Mayocardial infarction, NYHA Ⅳ heart failure | 1 year
  number of participants with death, mayocardial infarction or NYHA Ⅳ heart failure

SECONDARY OUTCOMES:
Slow reflow/no reflow | intraoperative
  number of participants with slow reflow/no reflow during PCI
Left ventricular function | 1 year
  left ventricular ejection fraction evaluated by ultrasound and MRI
Seattle Angina Questionnaire scores | 1 year
  Seattle Angina Questionnaire scores
Canadian Cardiovascular Society (CCS) Functional Angina classification | 1 year
  Canadian Cardiovascular Society (CCS) Functional Angina classification
6-minute walk distance (6MWD) | 1 year
  6-minute walk distance (6MWD)
Stroke | 1 year
  number of participants with stroke

CONTACTS AND LOCATIONS:
Overall Officials: Dongdong Sun, M.D.,Ph.D., Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China